CLINICAL TRIAL: NCT01381094
Title: Phase 2a Randomized, Double-Blind, Placebo-Controlled, Dose Range Study to Assess the Pharmacodynamic Response, Pharmacokinetics, Safety, and Tolerability of 42-Day Repeat Oral Doses of AKB-6548 in Subjects With Anemia Secondary to Chronic Kidney Disease (CKD), Stages 3 and 4
Brief Title: 42-Day Repeat Oral Dose Study of AKB-6548 in Participants With Chronic Kidney Disease and Anemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0005
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Results first posted 2022-07-01 (Actual); Last update posted 2022-07-01 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Kidney Disease
Keywords: anemia; chronic kidney disease; CKD; chronic renal insufficiency; renal impairment; erythropoietin; safety; efficacy; tolerability; pharmacokinetics
MeSH Terms: conditions — Anemia; Kidney Diseases; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- AKB-6548 240 mg (Experimental)
  Interventions: Drug: AKB-6548
- AKB-6548 370 mg (Experimental)
  Interventions: Drug: AKB-6548
- AKB-6548 500 mg (Experimental)
  Interventions: Drug: AKB-6548
- AKB-6548 630 mg (Experimental)
  Interventions: Drug: AKB-6548
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AKB-6548 — oral dose administered once daily for 42 days
  Arms: AKB-6548 240 mg; AKB-6548 370 mg; AKB-6548 500 mg; AKB-6548 630 mg
Drug: Placebo — oral Placebo administered once daily for 42 days
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the dose response (efficacy), pharmacodynamic response, pharmacokinetics, safety, and tolerability of orally administered AKB-6548 in pre-dialysis participants with anemia with repeat dosing for 42 days.

ELIGIBILITY:
Key Inclusion Criteria:

* 18 to 79 years of age, inclusive
* Chronic Kidney Disease (eGFR <60 mL/min), not yet on dialysis
* Hemoglobin (Hgb) ≤ 10.5 g/dL
* Transferring saturation ≥ 20%
* Ferritin ≥ 50 ng/mL

Key Exclusion Criteria:

* Body mass index >42
* Red blood cell transfusion within 12 weeks
* Androgen therapy within the previous 21 days prior to study dosing
* Therapy with any approved or experimental erythropoiesis stimulating agent (ESA) within the 11 weeks prior to the Screening visit
* Participants meeting the criteria of ESA resistance within the previous 4 months
* Individual doses of intravenous iron of greater than 250 mg within the past 21 days
* Aspartate aminotransferase or alanine aminotransferase >1.8x upper limit of normal (ULN)
* Alkaline phosphatase >2x ULN
* Total bilirubin >1.5x ULN
* Uncontrolled hypertension
* New York Heart Association Class III or IV congestive heart failure
* Myocardial infarction, acute coronary syndrome, or stroke within 6 months prior to dosing

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2011-06-15 (Actual); Primary Completion 2012-02-16 (Actual); Study Completion 2012-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (28):
- United States (28):
  - Pine Bluff, Arkansas
  - Covina, California
  - Los Angeles, California
  - Lynwood, California
  - Riverside, California
  - San Dimas, California
  - Whittier, California
  - Coral Springs, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Ocala, Florida
  - Augusta, Georgia
  - Macon, Georgia
  - Wichita, Kansas
  - Shreveport, Louisiana
  - Springfield, Massachusetts
  - Detroit, Michigan
  - Pontiac, Michigan
  - Warren, Michigan
  - Bethpage, New York
  - Mineola, New York
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Knoxville, Tennessee
  - Austin, Texas
  - Fort Worth, Texas
  - Houston, Texas
  - San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Martin ER, Smith MT, Maroni BJ, Zuraw QC, deGoma EM. Clinical Trial of Vadadustat in Patients with Anemia Secondary to Stage 3 or 4 Chronic Kidney Disease. Am J Nephrol. 2017;45(5):380-388. doi: 10.1159/000464476. Epub 2017 Mar 25. PMID 28343225

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 93 participants were enrolled and randomized into the study. Only 91 participants received the treatment.
Groups:
- AKB-6548 240 mg: Participants with anemia secondary to chronic kidney disease (CKD), stages 3 and 4 were administered with an oral dose of AKB-6548 240 milligrams (mg) capsule once daily (QD) for 42 days.
- AKB-6548 370 mg: Participants with anemia secondary to CKD, stages 3 and 4 were administered with an oral dose of AKB-6548 370 mg capsule QD for 42 days.
- AKB-6548 500 mg: Participants with anemia secondary to CKD, stages 3 and 4 were administered with an oral dose of AKB-6548 500 mg capsule QD for 42 days.
- AKB-6548 630 mg: Participants with anemia secondary to CKD, stages 3 and 4 were administered with an oral dose of AKB-6548 630 mg capsule QD for 42 days.
- Placebo: Participants with anemia secondary to CKD, stages 3 and 4 were administered with an oral dose of matching Placebo QD for 42 days.
Period: Overall Study
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Started | 18 | 18 | 17 | 19 | 19
Completed | 16 | 15 | 17 | 18 | 18
Not Completed | 2 | 3 | 0 | 1 | 1
Not completed — Adverse Event | 1 | 2 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal of informed consent | 0 | 1 | 0 | 0 | 0
Not completed — Participant given Aranesp injection | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population: All randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (12.17) | 68.9 (7.84) | 64.7 (9.47) | 64.9 (8.79) | 64.9 (9.97) | 65.5 (9.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 13 | 7 | 12 | 48
  Male | 9 | 11 | 4 | 12 | 7 | 43
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 4 | 4 | 4 | 5 | 24
  Not Hispanic or Latino | 11 | 14 | 13 | 15 | 14 | 67
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 0 | 0 | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1 | 2
  Black or African American | 6 | 4 | 4 | 7 | 3 | 24
  White | 10 | 13 | 13 | 9 | 14 | 59
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 1 | 4
CKD stage [Count of Participants; unit: Participants]
  Stage 3 | 5 | 4 | 4 | 5 | 5 | 23
  Stage 4 | 13 | 14 | 13 | 14 | 14 | 68

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change From Baseline in Hemoglobin (Hgb) to End of Treatment (Week 6)
Description: Absolute change from Baseline was calculated as the Week 6 (end of treatment) value minus the Baseline value. Baseline Hgb was defined as the average of the last two measurements obtained prior to dosing. If there was only one measurement prior to dosing, this measurement served as Baseline. A positive change from Baseline indicated that hemoglobin concentration increased.
Time Frame: Baseline, Week 6
Population: Modified intent-to-treat (MITT) population: All randomized participants who received at least one dose of study medication and had a Baseline (both Screening and Baseline for Hgb and red blood cells [RBC] count) and at least one post-baseline measurement. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (g/dL)
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Grams per deciliter (g/dL)
  Baseline | 9.46 (0.792) | 9.93 (0.643) | 9.86 (0.606) | 9.67 (0.796) | 9.83 (0.677)
  Change from Baseline at Week 6: number analyzed (Participants) | 16 | 15 | 17 | 18 | 18
  Change from Baseline at Week 6 | 0.77 (0.665) | 0.73 (0.623) | 1.25 (0.644) | 1.43 (0.668) | -0.03 (0.649)
Statistical Analysis 1: Comparison: AKB-6548 240 mg vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.80, 95% CI 2-sided [0.24 to 1.35]
Statistical Analysis 2: Comparison: AKB-6548 370 mg vs Placebo; Test type: Superiority; Mean Difference (Net) = 0.76, 95% CI 2-sided [0.20 to 1.33]
Statistical Analysis 3: Comparison: AKB-6548 500 mg vs Placebo; Test type: Superiority; Mean Difference (Net) = 1.28, 95% CI 2-sided [0.73 to 1.83]
Statistical Analysis 4: Comparison: AKB-6548 630 mg vs Placebo; Test type: Superiority; Mean Difference (Net) = 1.45, 95% CI 2-sided [0.91 to 2.00]
Statistical Analysis 5: Comparison: AKB-6548 240 mg vs AKB-6548 370 mg vs AKB-6548 500 mg vs AKB-6548 630 mg vs Placebo; Test type: Superiority; p < 0.0001, ANOVA

2. Secondary Outcome: Change From Baseline in Hgb at Week 1, Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline Hgb was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated that hemoglobin concentration increased.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
g/dL
  Baseline | 9.46 (0.792) | 9.93 (0.643) | 9.86 (0.606) | 9.67 (0.796) | 9.83 (0.677)
  Change from Baseline to Week 1: number analyzed (Participants) | 18 | 16 | 17 | 19 | 18
  Change from Baseline to Week 1 | 0.06 (0.559) | -0.12 (0.452) | 0.28 (0.439) | 0.29 (0.622) | 0.04 (0.531)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 16 | 18 | 19
  Change from Baseline to Week 2 | 0.16 (0.575) | 0.00 (0.590) | 0.54 (0.586) | 0.53 (0.455) | 0.14 (0.654)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 17 | 19 | 19
  Change from Baseline to Week 4 | 0.54 (0.659) | 0.36 (0.605) | 0.85 (0.650) | 1.06 (0.900) | 0.08 (0.613)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 17 | 18 | 18
  Change from Baseline to Week 6 | 0.77 (0.665) | 0.73 (0.623) | 1.25 (0.644) | 1.43 (0.668) | -0.03 (0.649)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 17 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | 0.78 (0.685) | 0.40 (0.553) | 1.04 (0.848) | 1.01 (0.872) | 0.06 (0.877)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.9355, 2 sided t-test/Wilcoxon Signed-rank Test; The comparison was made by using a 2-tailed, paired t-test (if the distribution was normal) or Wilcoxon Signed-Rank Test otherwise with an α=0.05
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.6594, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0203, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0369, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; Test type: Superiority — p-value was based on the comparison within treatment group (Change from Baseline to Week 1); p = 0.3713, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.1630, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.7615, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0040, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0003, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.3978, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0083, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0323, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0003, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.4230, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0023, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0009, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.5291, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0222, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9314, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

3. Secondary Outcome: Change From Baseline in Hematocrit (HCT) at Week 1, Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline HCT was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated HCT concentration increased.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells in blood
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 14 | 19 | 19
Percentage of red blood cells in blood
  Baseline | 29.0 (2.57) | 29.6 (2.45) | 30.4 (2.41) | 29.6 (3.68) | 29.8 (1.96)
  Change from Baseline to Week 1: number analyzed (Participants) | 18 | 16 | 14 | 19 | 18
  Change from Baseline to Week 1 | 0.5 (2.28) | 0.2 (1.87) | 1.2 (1.25) | 1.6 (2.65) | 0.2 (1.70)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 13 | 18 | 19
  Change from Baseline to Week 2 | 0.2 (2.46) | 0.1 (1.59) | 1.6 (2.33) | 1.5 (2.04) | 0.3 (2.06)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 14 | 19 | 19
  Change from Baseline to Week 4 | 1.7 (2.37) | 0.6 (1.67) | 3.1 (2.59) | 3.4 (3.52) | 0.1 (2.34)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 14 | 18 | 18
  Change from Baseline to Week 6 | 1.8 (2.71) | 2.1 (2.46) | 3.4 (2.47) | 4.3 (2.74) | -0.4 (2.40)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 14 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | 1.9 (2.30) | 0.7 (1.90) | 2.4 (2.62) | 2.8 (3.44) | 0.0 (2.78)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.5219, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.6743, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0078, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0301, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.4502, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.6967, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.7385, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0176, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0057, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.5551, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0086, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.2385, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0007, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.8895, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0127, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0076, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0007, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.5522, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0031, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.2188, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0054, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0037, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9521, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

4. Secondary Outcome: Change From Baseline in Red Blood Cell (RBC) Count at Week 1, Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline RBC count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated RBC count increased.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: 10^6 cells/microliter (10^6 cells/μL)
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
10^6 cells/microliter (10^6 cells/μL)
  Baseline | 3.21 (0.415) | 3.38 (0.286) | 3.37 (0.286) | 3.25 (0.366) | 3.34 (0.463)
  Change from Baseline to Week 1: number analyzed (Participants) | 18 | 16 | 17 | 19 | 18
  Change from Baseline to Week 1 | -0.01 (0.185) | -0.07 (0.178) | 0.09 (0.187) | 0.04 (0.227) | -0.02 (0.231)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 16 | 18 | 19
  Change from Baseline to Week 2 | 0.02 (0.183) | -0.05 (0.186) | 0.14 (0.229) | 0.11 (0.172) | 0.03 (0.281)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 17 | 19 | 19
  Change from Baseline to Week 4 | 0.16 (0.213) | 0.01 (0.202) | 0.26 (0.251) | 0.27 (0.294) | 0.02 (0.229)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 17 | 18 | 18
  Change from Baseline to Week 6 | 0.17 (0.243) | 0.18 (0.273) | 0.39 (0.252) | 0.41 (0.243) | -0.02 (0.223)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 17 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | 0.24 (0.242) | 0.06 (0.199) | 0.30 (0.248) | 0.26 (0.273) | 0.01 (0.290)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.3943, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.2096, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0637, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.5016, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.7549, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.5991, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.4258, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0336, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0258, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.2412, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0031, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.7705, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0024, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0006, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.6189, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0075, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0259, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.8898, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0010, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.2864, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0016, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9697, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

5. Secondary Outcome: Change From Baseline in Absolute Reticulocyte Count at Week 1, Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline Reticulocyte count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated reticulocyte count increased.
Time Frame: Baseline, Week 1, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 14 | 19 | 18
10^6 cells/μL
  Baseline | 0.0766 (0.02855) | 0.0569 (0.01891) | 0.0811 (0.01993) | 0.0674 (0.02715) | 0.0700 (0.03319)
  Change from Baseline to Week 1: number analyzed (Participants) | 18 | 16 | 14 | 19 | 17
  Change from Baseline to Week 1 | 0.0022 (0.01279) | 0.0134 (0.01733) | 0.0259 (0.02223) | 0.0289 (0.03152) | 0.0010 (0.01677)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 13 | 18 | 18
  Change from Baseline to Week 2 | 0.0012 (0.01505) | 0.0196 (0.01919) | 0.0346 (0.01997) | 0.0292 (0.01625) | -0.0015 (0.01091)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 14 | 19 | 18
  Change from Baseline to Week 4 | 0.0029 (0.01181) | 0.0128 (0.01586) | 0.0234 (0.02685) | 0.0206 (0.02369) | -0.0023 (0.01636)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 14 | 18 | 17
  Change from Baseline to Week 6 | -0.0020 (0.01736) | 0.0116 (0.02390) | 0.0061 (0.02217) | 0.0047 (0.02639) | -0.0004 (0.01788)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 16 | 13 | 14 | 17 | 15
  Change from Baseline to Follow-up Visit (up to Week 8) | -0.0042 (0.01900) | 0.0015 (0.02616) | -0.0152 (0.01467) | -0.0119 (0.02494) | -0.0035 (0.01522)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 1.0000, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0055, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0009, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 1); Test type: Superiority; p = 0.9722, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 1.0000, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0008, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.6579, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.4102, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0023, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0052, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0017, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.7378, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.3371, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0916, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.4656, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.1629, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.7032, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 21: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.5194, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 22: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.8516, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 23: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0017, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 24: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0656, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 25: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.6495, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Change From Baseline in Reticulocyte Hgb Content at Week 6
Description: Change from Baseline was calculated as the Week 6 value minus the Baseline value. Baseline Reticulocyte count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated reticulocyte Hgb content increased.
Time Frame: Baseline, Week 6
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Picogram
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 14 | 19 | 19
Picogram
  Baseline | 31.02 (2.945) | 31.44 (2.257) | 30.26 (2.605) | 31.54 (2.575) | 30.73 (2.634)
  Change From Baseline at Week 6: number analyzed (Participants) | 16 | 15 | 14 | 18 | 18
  Change From Baseline at Week 6 | 0.37 (0.971) | 0.29 (0.742) | 0.06 (0.964) | 0.15 (1.214) | 0.03 (1.104)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.2065, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.1807, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.7869, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.4743, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.6407, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Maximum Change From Baseline in Hgb
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline Hgb was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated that hemoglobin concentration increased.
Time Frame: Baseline; up to Week 8
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
g/dL
  Baseline | 9.46 (0.792) | 9.93 (0.643) | 9.86 (0.606) | 9.67 (0.796) | 9.83 (0.677)
  Maximum change from Baseline (up to Week 8) | 1.04 (0.585) | 0.82 (0.581) | 1.44 (0.675) | 1.54 (0.911) | 0.59 (0.568)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

8. Secondary Outcome: Maximum Change From Baseline in HCT
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline HCT was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated that HCT concentration increased.
Time Frame: Baseline; up to Week 8
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of red blood cells
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 14 | 19 | 19
Percentage of red blood cells
  Baseline | 29.0 (2.57) | 29.6 (2.45) | 30.4 (2.41) | 29.6 (3.68) | 29.8 (1.96)
  Maximum change from Baseline (up to Week 8) | 2.94 (2.578) | 2.56 (2.097) | 4.43 (2.277) | 4.84 (3.452) | 1.89 (1.729)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0004, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

9. Secondary Outcome: Maximum Change From Baseline in RBC Count
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline RBC Count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated that RBC count increased.
Time Frame: Baseline; up to Week 8
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
10^6 cells/μL
  Baseline | 3.21 (0.415) | 3.38 (0.286) | 3.37 (0.286) | 3.25 (0.366) | 3.34 (0.463)
  Maximum change from Baseline (up to Week 8) | 0.31 (0.210) | 0.22 (0.239) | 0.44 (0.249) | 0.44 (0.291) | 0.18 (0.183)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0043, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

10. Secondary Outcome: Maximum Change in Absolute Reticulocyte Count From Baseline
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline absolute reticulocyte count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline. A positive change from Baseline indicated that reticulocyte count increased.
Time Frame: Baseline; up to Week 8
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: 10^6 cells/μL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 14 | 19 | 18
10^6 cells/μL
  Baseline | 0.0766 (0.02855) | 0.0569 (0.01891) | 0.0811 (0.01993) | 0.0674 (0.02715) | 0.0700 (0.03319)
  Maximum Change from Baseline (up to Week 8) | 0.013 (0.0145) | 0.028 (0.0184) | 0.040 (0.0200) | 0.042 (0.0263) | 0.011 (0.0129)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0027, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group; Test type: Superiority; p = 0.0005, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

11. Secondary Outcome: Number of Participants With Absolute Change From Baseline in Hgb ≥ 0.4, 0.6, 0.8, and 1.0 g/dL at the End of Dosing Period
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline Hgb was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Up to Week 6 (End of the Dosing Period)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Participants
  Change from Baseline in Hgb ≥0.4 g/dL | 3 | 2 | 2 | 1 | 2
  Change from Baseline in Hgb ≥0.6 g/dL | 3 | 2 | 0 | 1 | 0
  Change from Baseline in Hgb ≥0.8 g/dL | 3 | 2 | 3 | 1 | 0
  Change from Baseline in Hgb ≥1.0 g/dL | 5 | 6 | 11 | 14 | 2

12. Secondary Outcome: Number of Participants With Change From Baseline in Hgb ≥5.0, 7.5, and 10.0% by the End of Dosing Period
Description: as for outcome 11
Time Frame: Up to Week 6 (End of The Dosing Period)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Participants
  % Change from Baseline in Hgb ≥5% | 4 | 3 | 1 | 1 | 2
  % Change from Baseline in Hgb ≥7.5% | 4 | 3 | 3 | 1 | 0
  % Change from Baseline in Hgb ≥10.0% | 5 | 5 | 11 | 14 | 2

13. Secondary Outcome: Number of Participants With Change From Baseline in HCT ≥5.0, 7.5, and 10.0% by the End of Dosing Period
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline HCT was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Up to Week 6 (End of The Dosing Period)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Participants
  % Change from Baseline in HCT ≥5% | 4 | 3 | 2 | 0 | 1
  % Change from Baseline in HCT ≥7.5% | 1 | 0 | 0 | 4 | 1
  % Change from Baseline in HCT ≥10.0% | 4 | 6 | 9 | 11 | 1

14. Secondary Outcome: Number of Participants With Change From Baseline in RBC Count ≥5.0, 7.5, and 10.0% by the End of Dosing Period
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline RBC Count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Up to Week 6 (End of The Dosing Period)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Participants
  % Change from Baseline in RBCs ≥5% | 4 | 3 | 2 | 3 | 1
  % Change from Baseline in RBCs ≥7.5% | 2 | 2 | 3 | 1 | 0
  % Change from Baseline in RBCs ≥10.0% | 2 | 4 | 8 | 11 | 1

15. Secondary Outcome: Number of Participants With Change From Baseline in Reticulocyte Count ≥6000, 12000, and 18000 Cells/uL by the End of Dosing Period
Description: Change from Baseline was calculated as the maximum value minus the Baseline value. Baseline reticulocytes count was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Up to Week 6 (End of The Dosing Period)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 17 | 19 | 19
Participants
  Change from Baseline in Reticulocytes ≥6000 cells/uL | 1 | 1 | 4 | 2 | 3
  Change from Baseline in Reticulocytes ≥12000 cells/uL | 1 | 3 | 0 | 3 | 1
  Change from Baseline in Reticulocytes ≥18000 cells/uL | 2 | 5 | 4 | 5 | 2

16. Secondary Outcome: Change From Baseline in Total Iron at Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline total iron was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Micrograms per deciliter (µg/dL)
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
Micrograms per deciliter (µg/dL)
  Baseline | 66.0 (18.68) | 77.8 (22.47) | 76.1 (32.01) | 60.7 (20.51) | 67.6 (21.12)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 14 | 18 | 19
  Change from Baseline to Week 2 | -1.8 (15.87) | -3.7 (18.96) | 10.9 (22.93) | 10.4 (24.54) | -4.1 (18.55)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 15 | 19 | 18
  Change from Baseline to Week 4 | -1.5 (21.62) | 4.0 (16.36) | -1.6 (20.49) | 13.2 (24.18) | -2.2 (20.47)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 15 | 18 | 18
  Change from Baseline to Week 6 | 3.6 (23.26) | 2.8 (15.44) | 3.7 (25.19) | 0.7 (16.54) | -8.6 (25.81)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 15 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | -7.4 (19.25) | -7.5 (22.90) | 0.9 (31.90) | 6.2 (18.50) | 3.4 (16.05)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.6051, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.5197, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.1073, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.1321, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.4358, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.8109, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.2575, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.8361, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0294, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.8809, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.4971, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.3994, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.5022, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.9916, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.2292, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.1331, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.5518, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9032, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.2387, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.4251, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

17. Secondary Outcome: Change From Baseline in Unsaturated Iron Binding Capacity at Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline Unsaturated Iron Binding Capacity was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
µg/dL
  Baseline | 153.4 (34.26) | 168.0 (52.46) | 173.1 (56.48) | 171.2 (38.77) | 175.5 (33.14)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 14 | 18 | 19
  Change from Baseline to Week 2 | 10.9 (18.78) | 22.4 (19.52) | 17.2 (32.16) | 21.3 (27.40) | -1.5 (20.61)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 15 | 19 | 18
  Change from Baseline to Week 4 | 14.4 (25.96) | 26.1 (22.30) | 31.5 (27.08) | 37.4 (20.16) | -3.7 (27.89)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 15 | 18 | 18
  Change from Baseline to Week 6 | 15.3 (30.52) | 34.0 (25.62) | 29.3 (16.06) | 49.6 (26.50) | -1.3 (17.81)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 15 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | 15.1 (30.46) | 16.2 (22.74) | -0.7 (23.06) | 3.9 (42.20) | 0.7 (20.72)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0448, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0004, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0813, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0038, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.6861, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0553, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0004, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.7379, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0720, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.6781, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0524, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0367, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.6671, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.6861, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9012, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

18. Secondary Outcome: Change From Baseline in Iron Saturation at Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline iron saturation was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Percentage of saturation
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
Percentage of saturation
  Baseline | 30.4 (7.56) | 32.4 (9.82) | 31.4 (13.35) | 26.5 (10.17) | 27.7 (6.60)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 14 | 18 | 19
  Change from Baseline to Week 2 | -1.5 (6.26) | -3.8 (7.34) | 1.4 (9.15) | 0.6 (8.81) | -0.9 (7.86)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 15 | 19 | 18
  Change from Baseline to Week 4 | -1.9 (8.10) | -2.3 (7.00) | -3.7 (7.91) | -0.2 (6.52) | -0.2 (8.65)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 15 | 18 | 18
  Change from Baseline to Week 6 | -0.3 (9.24) | -3.8 (6.36) | -2.3 (7.69) | -4.6 (6.44) | -2.1 (9.09)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 15 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | -4.1 (7.08) | -3.9 (8.90) | 0.5 (9.94) | 1.6 (9.27) | 1.2 (5.80)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.3953, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0850, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.6045, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.7743, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.5326, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.3465, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.2756, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.1414, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.6941, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.9403, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.8310, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0654, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.4169, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0103, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.3968, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0325, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.2151, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.8436, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.5962, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.3957, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

19. Secondary Outcome: Change From Baseline in Total Iron Binding Capacity (TIBC) at Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline TIBC was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6, Follow-up Visit (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: µg/dL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
µg/dL
  Baseline | 219.4 (39.39) | 245.8 (54.61) | 249.2 (45.29) | 231.8 (36.19) | 243.1 (40.02)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 14 | 18 | 19
  Change from Baseline to Week 2 | 9.2 (16.34) | 18.7 (18.09) | 28.1 (22.32) | 31.7 (28.73) | -5.5 (22.51)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 15 | 19 | 18
  Change from Baseline to Week 4 | 12.9 (24.97) | 30.1 (16.20) | 29.9 (24.08) | 50.5 (28.64) | -5.9 (17.96)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 15 | 18 | 18
  Change from Baseline to Week 6 | 18.8 (28.81) | 36.8 (27.76) | 33.0 (28.54) | 50.3 (27.80) | -9.9 (25.70)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 15 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | 7.8 (34.88) | 8.7 (18.15) | 0.2 (25.82) | 10.2 (30.15) | 4.1 (23.83)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0294, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0021, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0004, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0925, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0433, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0005, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.1626, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0366, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0004, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0012, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.1779, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.5867, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.1306, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.9889, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.2026, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.5703, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

20. Secondary Outcome: Change From Baseline in Ferritin at Week 2, Week 4, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline ferritin was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 4, Week 6, Follow-up (up to Week 8)
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
Nanograms per milliliter (ng/mL)
  Baseline | 349.5 (226.27) | 245.8 (215.18) | 332.3 (330.81) | 240.2 (142.10) | 200.8 (115.99)
  Change from Baseline to Week 2: number analyzed (Participants) | 16 | 16 | 14 | 18 | 19
  Change from Baseline to Week 2 | -66.0 (67.72) | -41.7 (53.18) | -72.0 (75.89) | -58.9 (54.72) | -12.9 (35.49)
  Change from Baseline to Week 4: number analyzed (Participants) | 17 | 16 | 15 | 19 | 19
  Change from Baseline to Week 4 | -69.8 (101.67) | -48.7 (63.08) | -89.6 (138.80) | -80.6 (64.50) | -20.5 (39.24)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 15 | 18 | 18
  Change from Baseline to Week 6 | -65.5 (115.89) | -59.4 (58.76) | -88.9 (64.66) | -86.6 (62.73) | -19.6 (41.72)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 17 | 14 | 15 | 17 | 16
  Change from Baseline to Follow-up Visit (up to Week 8) | -50.4 (91.22) | -37.7 (73.31) | -86.1 (67.75) | -27.4 (107.42) | -20.2 (39.35)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0092, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.0012, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 2); Test type: Superiority; p = 0.1157, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 6: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0069, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 7: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0034, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 8: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0067, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 9: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 10: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 4); Test type: Superiority; p = 0.0401, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 11: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0042, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 12: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 13: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0002, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 14: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 15: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Week 6); Test type: Superiority; p = 0.0422, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 16: Comparison: AKB-6548 240 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0232, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 17: Comparison: AKB-6548 370 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0243, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 18: Comparison: AKB-6548 500 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 19: Comparison: AKB-6548 630 mg; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.1089, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 20: Comparison: Placebo; p-value was based on the comparison within treatment group (Change from Baseline to Follow-up); Test type: Superiority; p = 0.0833, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

21. Secondary Outcome: Change From Baseline in Erythropoietin at Week 2, Week 6, and Follow-up Visit (up to Week 8)
Description: Change from Baseline was calculated as the visit value minus the Baseline value. Baseline erythropoietin was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 2, Week 6, Follow-up Visit (up to Week 8)
Population: Intent-to-treat (ITT) population: All randomized participants who received at least one dose of study medication. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 15 | 19 | 19
ng/mL
  Baseline | 18.011 (56.3608) | 4.339 (4.1462) | 7.287 (8.8333) | 8.826 (10.2773) | 6.963 (14.1425)
  Change from Baseline to Week 2: number analyzed (Participants) | 17 | 16 | 13 | 18 | 19
  Change from Baseline to Week 2 | -3.538 (20.3172) | 0.606 (3.2070) | 1.142 (11.8961) | -2.483 (9.5483) | -0.850 (9.3370)
  Change from Baseline to Week 6: number analyzed (Participants) | 16 | 15 | 14 | 18 | 18
  Change from Baseline to Week 6 | -3.050 (15.1756) | -1.013 (3.9836) | -3.329 (5.9821) | -0.372 (14.4615) | -1.492 (10.1597)
  Change from Baseline to Follow-up Visit (up to Week 8): number analyzed (Participants) | 16 | 12 | 14 | 17 | 15
  Change from Baseline to Follow-up Visit (up to Week 8) | -3.853 (15.1335) | -0.563 (5.5372) | -2.061 (6.2689) | -4.844 (9.4601) | -2.650 (8.2146)

22. Secondary Outcome: Change From Baseline in Hepcidin at Week 6
Description: Change from Baseline was calculated as the Week 6 value minus the Baseline value. Baseline hepcidin was defined as the average of the last two measurements obtained prior to dosing; if there was only one value prior to dosing, this value served as Baseline.
Time Frame: Baseline, Week 6
Population: MITT population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 16 | 15 | 19 | 19
ng/mL
  Baseline | 326.35 (222.037) | 241.03 (158.871) | 242.51 (117.326) | 282.75 (239.266) | 258.29 (144.115)
  Change from Baseline at Week 6 | -28.64 (185.263) | -90.91 (106.826) | -85.01 (45.864) | -144.90 (184.640) | -32.54 (103.937)
Statistical Analysis 1: Comparison: AKB-6548 240 mg; Test type: Superiority; p = 0.5456, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: AKB-6548 370 mg; Test type: Superiority; p = 0.0053, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: AKB-6548 500 mg; Test type: Superiority; p < 0.0001, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 4: Comparison: AKB-6548 630 mg; Test type: Superiority; p = 0.0040, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]
Statistical Analysis 5: Comparison: Placebo; Test type: Superiority; p = 0.2017, 2 sided t-test/Wilcoxon Signed-rank Test; [statistical method as in outcome 2, analysis 1]

23. Secondary Outcome: Mean Plasma Vadadustat Concentrations on Week 2 and Week 4
Description: Plasma samples were collected for the analysis.
Time Frame: Week 2: Pre-dose and post-dose; Week 4: Pre-dose
Population: Pharmacokinetic (PK) Population: All participants in the ITT population that had pre-dose PK sampling that fell within a range of 18 to 30 hours after the previous dose of study medication or post-dose PK sampling that fell in a range of 2 to 8 hours post-dose. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg
Number analyzed (Participants) | 17 | 16 | 16 | 18
μg/mL
  Week 2 Pre-Dose: number analyzed (Participants) | 16 | 15 | 16 | 18
  Week 2 Pre-Dose | 4358.28 (2549.623) | 6640.04 (5141.484) | 10791.79 (9823.143) | 12443.17 (17095.495)
  Week 2 Post-Dose: number analyzed (Participants) | 17 | 16 | 15 | 18
  Week 2 Post-Dose | 17036.82 (8035.308) | 21371.63 (8664.304) | 39892.00 (19891.284) | 41656.11 (20002.713)
  Week 4 Pre-Dose: number analyzed (Participants) | 16 | 16 | 15 | 18
  Week 4 Pre-Dose | 4698.21 (3520.520) | 7884.56 (5517.132) | 14274.80 (16141.439) | 17700.17 (19532.648)

24. Secondary Outcome: Mean Plasma Vadadustat Acyl-Glucuronide Concentrations on Week 2 and Week 4
Description: Plasma samples were collected for the analysis.
Time Frame: Week 2: Pre-dose; Week 4: Pre-dose
Population: PK population. Participants with available data were included in the analysis.
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg
Number analyzed (Participants) | 15 | 15 | 13 | 16
μg/mL
  Week 2 Pre-Dose: number analyzed (Participants) | 15 | 12 | 13 | 16
  Week 2 Pre-Dose | 1848.4 (979.73) | 2708.5 (1879.02) | 5900.1 (8309.24) | 6425.0 (7214.67)
  Week 4 Pre-Dose: number analyzed (Participants) | 13 | 15 | 13 | 14
  Week 4 Pre-Dose | 1999.3 (1427.74) | 2687.5 (2027.63) | 6866.9 (9247.39) | 7960.8 (6643.98)

25. Secondary Outcome: Number of Participants Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Description: An adverse event (AE) was defined as any untoward medical occurrence (including a clinically significant abnormal laboratory finding) that occurred in the protocol-specified AE reporting period. A TEAE included medical conditions, signs, and symptoms not previously observed in the participant that emerged during the protocol-specified AE reporting period, including signs or symptoms associated with pre-existing underlying conditions that were not present prior to the AE reporting period. A SAE included AEs that met one or more of the following criteria/outcomes: death, life-threatening, in-patient hospitalization or prolongation of existing hospitalization, persistent or significant disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Up to Week 8 (Follow-up Visit 2 weeks after last dose)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19
Participants
  TEAEs | 9 | 6 | 8 | 11 | 11
  SAEs | 2 | 3 | 1 | 1 | 1

26. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Vital Signs Parameter
Description: Parameters assessed for vital signs included sitting blood pressure, pulse, respiratory rate, and body temperature. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Week 8 (Follow-up Visit 2 weeks after last dose)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19
Participants | 0 | 0 | 0 | 0 | 0

27. Secondary Outcome: Number of Participants With Clinically Significant Abnormal 12-Electrocardiogram (ECG) Findings
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. Clinical significance is determined by the investigator. The investigator was responsible for reviewing laboratory results for clinical significance.
Time Frame: Up to Week 8 (Follow-up Visit 2 weeks after last dose)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19
Participants | 0 | 0 | 0 | 0 | 0

28. Secondary Outcome: Mean Change From Baseline in PR Interval, QT Interval, QRS Interval, and QT Corrected (QTc) Interval
Description: A standard 12-lead ECG was performed following dosing in a supine position for approximately 10 minutes. ECGs were taken prior to blood draws when possible. The parameters evaluated from the participant ECG trace included PR interval, QT interval, QRS interval, and QTc (corrected).
Time Frame: Baseline, Week 6
Population: ITT population.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19
Milliseconds
  Baseline PR Interval: number analyzed (Participants) | 18 | 17 | 16 | 17 | 18
  Baseline PR Interval | 156.7 (46.90) | 174.6 (40.89) | 172.8 (51.06) | 187.8 (45.72) | 175.8 (31.82)
  Change from Baseline PR Interval: number analyzed (Participants) | 17 | 18 | 17 | 19 | 19
  Change from Baseline PR Interval | -0.8 (22.95) | 2.2 (12.37) | 11.4 (29.72) | -11.7 (63.75) | -0.4 (13.07)
  Baseline QRS Duration | 94.9 (21.35) | 113.8 (37.57) | 97.1 (28.07) | 94.5 (12.65) | 94.6 (12.52)
  Change from Baseline QRS Duration: number analyzed (Participants) | 18 | 15 | 16 | 19 | 18
  Change from Baseline QRS Duration | 4.1 (9.52) | 2.0 (13.29) | -1.3 (7.23) | 1.4 (10.28) | -1.6 (5.33)
  Baseline QT Interval | 412.0 (41.59) | 421.4 (46.58) | 419.0 (44.97) | 406.9 (42.97) | 419.1 (40.10)
  Change from Baseline QT Interval: number analyzed (Participants) | 18 | 15 | 16 | 19 | 18
  Change from Baseline QT Interval | 3.8 (24.78) | 7.8 (25.33) | -1.6 (19.83) | 4.5 (24.10) | 11.0 (23.35)
  Baseline QTC Interval | 424.9 (27.70) | 436.3 (37.56) | 445.1 (36.10) | 427.6 (23.60) | 435.6 (17.90)
  Change from Baseline QTC Interval: number analyzed (Participants) | 18 | 15 | 16 | 19 | 18
  Change from Baseline QTC Interval | 5.1 (14.33) | 3.6 (17.65) | -5.8 (20.70) | -1.6 (16.74) | 3.3 (21.46)

29. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Parameter Values
Description: Parameters assessed for laboratory values included hematology, serum chemistry, C-reactive protein, DHEA-S, VEGF, and cystatin C. The investigator was responsible for reviewing laboratory results for clinically significant changes.
Time Frame: Up to Week 8 (Follow-up Visit 2 weeks after last dose)
Population: ITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
Number analyzed (Participants) | 18 | 18 | 17 | 19 | 19
Participants | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to Week 8 (Follow-up Visit 2 weeks after last dose)
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported.
Arm/Group | AKB-6548 240 mg | AKB-6548 370 mg | AKB-6548 500 mg | AKB-6548 630 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 1/18 | 0/17 | 0/19 | 0/19
Serious Adverse Events (participants affected / at risk) | 2/18 | 3/18 | 1/17 | 1/19 | 1/19
Other Adverse Events (participants affected / at risk) | 9/18 | 5/18 | 8/17 | 11/19 | 11/19
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AKB-6548 240 mg (N=18) | AKB-6548 370 mg (N=18) | AKB-6548 500 mg (N=17) | AKB-6548 630 mg (N=19) | Placebo (N=19)
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Azotaemia (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Cardiac pacemaker replacement (Cardiac disorders) | 1 | 0 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AKB-6548 240 mg (N=18) | AKB-6548 370 mg (N=18) | AKB-6548 500 mg (N=17) | AKB-6548 630 mg (N=19) | Placebo (N=19)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 2
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 1 | 0
Ear haemorrhage (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 2 | 1 | 2
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Adverse drug reaction (General disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1 | 0 | 1
Pain (General disorders) | 0 | 0 | 0 | 0 | 1
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 2 | 0 | 1 | 1 | 0
Viral infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Wound infection pseudomonas (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Joint sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Blood bicarbonate decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood glucose decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0 | 0 | 0
Transferrin saturation decreased (Investigations) | 0 | 0 | 0 | 1 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 3 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1
Vitamin d deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Hair texture abnormal (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2 | 3
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No